CLINICAL TRIAL: NCT06313073
Title: Neoadjuvant Radiotherapy Versus Adjuvant Radiotherapy for Breast Cancer: A Phase II Exploratory Randomized Controlled Clinical Study
Brief Title: Neoadjuvant Radiotherapy for Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Director, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHFL-BC-01
Record Dates: First submitted 2024-02-26; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Neoadjuvant Radiotherapy; Breast Cancer
Keywords: neoadjuvant radiotherapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy; Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant radiotherapy (Experimental): The patient received synchronous radiotherapy and chemotherapy before surgery. CTV : 40Gy/15fx/3w, sequential GTV： 8.7-10Gy/3-4 Fx.
  Interventions: Radiation: Neoadjuvant radiotherapy
- Adjuvant radiotherapy (Active Comparator): The patient underwent postoperative adjuvant radiotherapy. CTV : 40Gy/15fx/3w, sequential GTV： 8.7-10Gy/3-4 Fx.
  Interventions: Radiation: adjuvant radiotherapy

INTERVENTIONS:
Radiation: Neoadjuvant radiotherapy — The patient received synchronous radiotherapy and chemotherapy before surgery. CTV : 40Gy/15fx/3w, sequential GTV： 8.7-10Gy/3-4 Fx.CTV : 40Gy/15fx/3w, sequential GTV： 8.7-10Gy/3-4 Fx.
  Arms: Neoadjuvant radiotherapy
Radiation: adjuvant radiotherapy — The patient received radiotherapy after surgery. CTV : 40Gy/15fx/3w, sequential GTV： 8.7-10Gy/3-4 Fx.CTV : 40Gy/15fx/3w, sequential GTV： 8.7-10Gy/3-4 Fx.
  Arms: Adjuvant radiotherapy

SUMMARY:
The goal of this clinical trial is to compare the effects of neoadjuvant radiotherapy and adjuvant radiotherapy in patients with breast cancer.

The main questions it aims to answer are:

* The clinical effect of neoadjuvant radiotherapy for breast cancer was determined according to the postoperative specimens.
* Evaluate the acute and late toxicity of preoperative radiotherapy Participants will be randomly divided into two groups: the neoadjuvant radiotherapy group and the adjuvant radiotherapy group.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Age range from 18 to 70 years old;
* The pathological diagnosis is invasive cancer, and immunohistochemical examination has been performed to confirm the status of ER, PR, HER2, Ki67, etc;
* Clarify the BRCA gene mutation status;
* Patients who have a baseline stage of T1-3N0-3M0 and meet one of the following conditions and require neoadjuvant therapy: ① mass>5cm; ② Axillary lymph node metastasis; ③ HER-2 positive; ④ Three Yin type; ⑤ Those who have a desire to preserve breast, but have a large ratio of tumor size to breast volume, making it difficult to preserve breast;
* Baseline estimation requires adjuvant radiotherapy, which meets one of the following conditions: ① performing breast conserving surgery; ② T3 or N positive patients after mastectomy and axillary dissection; ③ After mastectomy, sentinel lymph nodes were positive and axillary dissection was not performed;
* KPS score ≥ 80;
* The tumor must be visible in CT scan;
* Patients must undergo magnetic resonance imaging to help determine the contour of the tumor and exclude other lesions. If other lesions are found, biopsy must be performed on these lesions and the result is negative before continuing treatment;
* No history of serious internal medicine diseases or other serious comorbidities, such as a history of mental illness, allergies, etc;
* Sign an informed consent form.

Exclusion Criteria:

* Clinical or pathological stage T4 or M1 breast cancer;
* Received preoperative neoadjuvant therapy;
* Pathological confirmation shows that there is no invasive cancer component in DCIS;
* Double breast cancer or previous contralateral breast cancer;
* Imaging examination suggests suspicious malignant lesions in the ipsilateral or contralateral breast, which have not been pathologically confirmed to be benign;
* KPS score ≤ 70;
* There is active infection currently;
* Concomitant with severe heart, liver, kidney, hematopoietic and neurological diseases, psychiatric patients, or estimated survival time<6 months;
* History of malignant tumors in other areas, excluding curable non melanoma skin cancer and cervical cancer in situ;
* History of radiation therapy at the site of previous radiation therapy;
* Pregnancy and lactation period;
* Those with poor compliance or life-threatening conditions who cannot complete treatment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
pCR | up to 3 weeks
  pathological complete remission

SECONDARY OUTCOMES:
RCB | up to 3 weeks
  residual cancer burden

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No